CLINICAL TRIAL: NCT02325492
Title: Medical Dissolution of Cholesterol Gallstones Using Oral Aramchol - A Proof of Concept Phase IIa Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol redesign
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aramchol006
Record Dates: First submitted 2014-11-12; First posted 2014-12-25 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2014-12

CONDITIONS: Gallstones
Keywords: bariatric surgery; NASH; ARAMCHOL
MeSH Terms: conditions — Gallstones | interventions — aramchol; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aramchol 400 mg (Experimental): • One tablet of Aramchol 400 mg and one tablet of Placebo
  Interventions: Drug: Aramchol; Drug: Placebo; Device: Ultrasound
- Aramchol 600 mg (Experimental): • One tablet of Aramchol 400 mg and one tablet of Aramchol 200 mg.
  Interventions: Drug: Aramchol; Device: Ultrasound
- Placebo (Placebo Comparator): • Two tablet of Aramchol matching placebo.
  Interventions: Drug: Placebo; Device: Ultrasound

INTERVENTIONS:
Drug: Aramchol
  Arms: Aramchol 400 mg; Aramchol 600 mg
Drug: Placebo
  Arms: Aramchol 400 mg; Placebo
Device: Ultrasound

SUMMARY:
This is a one center, Phase IIa, randomized, double blind, placebo controlled study designed to evaluate the efficacy and safety of two Aramchol doses in subjects 18 to 75 years of age, with newly formed cholesterol gallstones in their gallbladder following bariatric surgery confirmed by gallbladder ultrasound ..

DETAILED DESCRIPTION:
This is a one center, Phase IIa, randomized, double blind, placebo controlled study designed to evaluate the efficacy and safety of two Aramchol doses in subjects 18 to 75 years of age, with newly formed cholesterol gallstones in their gallbladder following bariatric surgery confirmed by gallbladder ultrasound performed in a period of 3 & 6 months following surgery before entering the study. All patients have ultrasonography evidence of clear gallbladder before the bariatric surgery.

Eligible subjects will be enrolled into three treatments arms: Aramchol 400 mg and 600 mg tablets and placebo tablets in ratio 1:1:1.

The subjects will be evaluated at study sites for 6 scheduled visits: at weeks -4 - 0 screening visit, Day 0 - baseline, weeks 2, 4, 8& 12 (Termination/early termination visit).

During the screening period the presence and number of cholesterol gallstones will be evaluated by gallbladder Ultrasound.

During the study the following assessments will be performed:

* Vital signs will be measured at each study visit.
* A physical examination will be performed at the screening visit, and termination/early termination visit.
* The following safety blood tests will be performed: complete blood count (CBC), serum chemistry (including electrolytes, liver enzymes, direct and total bilirubin, glucose, HbA1C, lipid profile which include cholesterol, HDL, LDL and VLDL, CPK, creatinine, urea, albumin, alkaline phosphatase), coagulation (fibrinogen, PT/INR, aPTT), ESR and urinalysis during the screening visit, baseline, week 2, 4, 8 and 12 (termination/early termination) visits. Serology (HBV, HCV and HIV) will be performed during the screening visit. β-hCG in women of child bearing potential will be performed during the screening visit.
* Body weight will be measured in screening, baseline and end of treatment visits. Height will be measured during the screening visit.
* ECG will be performed during the screening and end of treatment visits.
* Blood for Metabolomics will be collected at baseline and end of treatment visits.
* Ultrasound will be performed at screening visit, baseline, week 4, 8 and termination/early termination visits.
* Adverse events will be monitored throughout the study.
* Concomitant Medications will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 to 75 years.
2. Presence of newly formed gallstones (size up to 6 mm) with or without sludge diagnosed by ultrasound within 3 or 6 months after bariatric surgery following normal ultrasound.
3. Bariatric surgery conducted during the last 12 months
4. Patients with "sleeve gastrectomy" or laparoscopic banding of the upper stomach will be included.
5. Signature of the written informed consent.
6. Negative pregnancy test at study entry for females of child bearing potential.
7. Females of child bearing potential practicing reliable contraception throughout the study period (not including oral contraceptives).
8. Hypertensive patients must be well controlled by stable dose of anti-hypertensive medication for at least 2 months prior to screening (and the stable dose can be maintained throughout the study).
9. Patients treated with vitamin E(>400IU/die), or Polyunsaturated fatty acid (>2g/d) or Ursodeoxycholic acid or fish oil can be included if drugs are stopped at least 3 months prior to study enrollment to the study and up to it end.
10. For patients with type 2 Diabetes, glycaemia must be controlled (Glycosylated Hemoglobin A1C ≤ 8% while any HbA1C increment should not exceed 1% during 6 month prior to enrollment). If glycaemia is controlled by medications, qualitative change is not permitted within 3 months prior to randomization and should be avoided during the study. Treatments with Metformin, Sulfamides and Insulin are authorized. Sulfamides and insulin are permitted if glycaemia is self-monitored by the patient.

Exclusion Criteria:

1. Patients with ultrasonography evidence of gallstones in gallbladder before having the bariatric surgery.
2. Patients with no clear ultrasonography evidence of gallstones -free gallbladder during the year prior their bariatric surgery.
3. Patients with ultrasonography evidence of gallstones more than 1 year following bariatric surgery.
4. Patients with ultrasonography evidence of gallstones in size greater than 9 mm less than 1 year following bariatric surgery.
5. Weight >140 Kg or BMI >40
6. Known alcohol and/or any other drug abuse or dependence in the last five years
7. Known history or presence of clinically significant cardiovascular, hepatic, gastrointestinal, neurologic, pulmonary, endocrine, psychiatric, neoplastic disorder or nephritic syndrome.
8. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs including bile salt metabolism (e.g. inflammatory bowel disease (IDB); previous intestinal (ileal or colonic) operation; chronic pancreatic; celiac disease or previous vagotomy
9. Uncontrolled blood pressure
10. Patients with HIV
11. Patients with renal dysfunction eGFR< 60.
12. Patients with pancreatitis, cholangitis or cholecystitis in the previous 4 months.
13. Women who are pregnant or breastfeeding
14. Type 1 Diabetes.
15. .Metformin, Fibrates, Statins, Insulin, Sulfonilurea not provided on a stable dose in the last 6 months.
16. Patients who are treated with Valproic acid, Tamoxifen, Methotreksate, Amiodaron.
17. Treatment with Rifaximin.
18. Homeopathic and/or Alternative treatments. Any treatment should be stopped before the screening period.
19. Serum creatine phosphokinase (CPK), ALT, AST and/or alkaline phosphatase >3X the upper limit of normal (ULN). Patients with an intermittent CPK elevation may have the repeated measurement prior to randomization; a CPK retest > 3X ULN leads to exclusion.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Complete dissolution of existing gallstones proven by repeated US examined gallbladder | At baseline and week 12
  Change from baseline measured by US scan

SECONDARY OUTCOMES:
Decrease of more than a 50% in number of stones. (change from baseline) | At baseline and week 12
  change from baseline measured by US scan
Prevention of formation of new gallstones during the study period | At baseline and week 12
  change from baseline measured by US scan
Dissolution of sludge. | At baseline and week 12
  change from baseline measured by US scan

CONTACTS AND LOCATIONS:
Overall Officials: Asnat Raziel, MD, Principal Investigator — Assuta Medical Center
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel